CLINICAL TRIAL: NCT03051880
Title: The Preventive Effect of Topical EGF Cream for Dermatologic Adverse Events Related to EGFR Inhibitors
Brief Title: Preventive Effect of EGF Cream for Cutaneous Adverse Event of EGFR Inhibitors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jung Min Bae, Clinical Assistant Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VC16EISE0180
Record Dates: First submitted 2016-12-02; First posted 2017-02-14 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Drug-Related Side Effects and Adverse Reactions; Epidermal Growth Factor
Keywords: Epidermal Growth Factor
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Repair Control EGF® (Experimental): EGF cream was applied. One half side of face and one hand were treated with emollient containing EGF.
  Interventions: Drug: Repair Control EGF®
- Cream without rhEGF (Placebo Comparator): Placebo cream without EGF was applied. The other half side of face and the other hand were treated with only emollient which was not containing EGF.
  Interventions: Drug: Cream without rhEGF

INTERVENTIONS:
Drug: Repair Control EGF® — A Split face study was done. Patients applied 1 finger tip unit of EGF cream on one side of face, twice a day for 8 weeks. Also, to evaluate the preventive effect of paronychia, patients applied same cream on the finger tips of one side hand, twice a day for 8 weeks.
  EGF cream(Repair Control EGF®) containing 10 ppm of rhEGF was prepared at D.N. Co., Ltd. (Seoul, South Korea)
  Other Names: EGF cream containing 10 ppm of rhEGF
  Arms: Repair Control EGF®
Drug: Cream without rhEGF — A Split face study was done. Patients applied 1 finger tip unit of cream on the other side of face, twice a day for 8 weeks. Patients applied same cream on the finger tips of the other side hand, twice a day for 8 weeks.
  Placebo cream was prepared at at D.N. Co., Ltd. (Seoul, South Korea), consisted of same ingredient with EGF cream except rhEGF
  Arms: Cream without rhEGF

SUMMARY:
The purpose of this study is to evaluate the preventive efficacy of topical EGF cream for dermatologic adverse events related to EGFR inhibitors.

DETAILED DESCRIPTION:
Epidermal growth factor receptor(EGFR) is involved in cell proliferation and is overexpressed or abnormally activated in malignant tumors originating from the colon, breast, ovary, pancreas, and lung. EGFR tyrosine kinase inhibitor(TKI), gefitinib, erlotinib, and afatinib have been for the treatment of cancer associated with EGFR gene mutation. In addition, monoclonal antibodies to EGFR, such as cetuximab and panitumumab, have been used as a chemotherapy for rectal cancer without ras gene mutation and advanced head and neck cancer.

The incidence of cutaneous toxicity of EGFR inhibitors is reported to be 75-80%. Clinical features include acneform folliculitis, xerosis, paronychia, and itching. Of these, about 10% of patients with Grade 3 or greater have a detrimental effect on quality of life and adherence to treatment, resulting in impaired therapeutic results.

There have been many attempts to prevent or treat such skin toxicity. However, there has been no scientifically proven treatment until now.

There is a growing interest in the role of EGF emulsifiers in the treatment of skin adverse effects of EGFR inhibitors, as a result of studies that improve acne significantly compared to placebo.

The purpose of this study is to evaluate the preventive efficacy of EGF cream in the treatment of skin adverse effects in patients with malignant tumors treated with EGFR inhibitor (TKI or monoclonal antibody).

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years old
* Patients scheduled to receive EGFR inhibitors (gefitinib, erlotinib, afatinib, cetuximab, etc.) as malignant tumors
* Patients who can understand and follow the protocol
* Patients who spontaneously agreed to the study

Exclusion Criteria:

* Patients with a history of antibiotic treatment, local and systemic steroid therapy within 4 weeks of other skin disorders
* Patients with existing acne history
* Breastfeeding or pregnant women
* Patients who are deemed unsuitable for the examination by the researcher's judgment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The change of acneiform eruption caused by use of EGFR inhibitor | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  To evaluate the development and severity of acneiform eruption, the investigators take a photograph of full face and hands on every visit.
  If the acneiform eruption develop, the severity will be assessed based on the Korean Acne Grading System(KAGS).

SECONDARY OUTCOMES:
the change paronychia caused by use of EGFR inhibitor | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  The paronychia lesion will be assessed by CTCAE.
the change of skin hydration | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  It measured with Corneometer® (CM820/825, C-K Electronics, Cologne, Germany). It shows in arbitrary units(AU) and the unit is from 0 to 220.
the change of sebum production | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  It measured with Sebumeter® (SM815; C-K Electronics, Cologne, Germany). It is measured at forehead, cheek and chin, presented as /㎍ ㎠. It shows in arbitrary units(AU) and the unit is from 0 to 220.
Investigator's global assessment score | Baseline, 8 weeks
  Investigator's global assessment (IGA) Score will be assessed with 5-point scale (-1 = worsen to 3 =marked improvement).
Patient's global assessment score | Baseline, 8 weeks
  Patient's global assessment (PGA) score will be assessed with a 5-point scale (-1 = worsen, to 3 = marked improvement).
The side effects of product | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  It will be assessed by patient-report.
  - Any event developed during the trials can be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Min B, MD, PhD, Study Chair — The Catholic University of Korea
Locations (1):
- St. Vincent's Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided